CLINICAL TRIAL: NCT06096779
Title: A Phase II, Open-label, Multi-cohort, Multicenter Study in Patients With Unresectable Hepatocellular Carcinoma and Child-pugh B7 and B8 Cirrhosis
Brief Title: A Study Evaluating Atezolizumab, With or Without Bevacizumab, in Participants With Unresectable Hepatocellular Carcinoma and Child-pugh B7 and B8 Cirrhosis
Acronym: Kirros
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML44719
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Cirrhosis; Liver Cancer; Liver Tumor; Child-pugh B; Hepatocellular Carcinoma; Atezolizumab; Bevacizumab; Immune Checkpoint Inhibitor; Digestive System Neoplasms; Kirros; ML44719; Liver Disease; Genentech; Immunotherapy; CPB; CPB 7; CPB 8; Tecentriq; Avastin; HCC; Cirrhotic Liver; Fatty Liver
MeSH Terms: conditions — Carcinoma, Hepatocellular; Fibrosis; Liver Neoplasms; Digestive System Neoplasms; Liver Diseases; Fatty Liver | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: Atezolizumab+Bevacizumab (Experimental): Participants will receive atezolizumab plus bevacizumab until unacceptable toxicity or loss of clinical benefit, as determined by the investigator.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab
- Cohort B: Atezolizumab (Experimental): Participants will receive atezolizumab until unacceptable toxicity or loss of clinical benefit, as determined by the investigator.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered at a dose of 1200 milligrams (mg) by intravenous (IV) infusion on Day 1 of each 21-day cycle.
  Other Names: Tecentriq; RO5541267
Drug: Bevacizumab — Bevacizumab will be administered at a dose of 15 milligrams per kilogram (mg/kg) by IV infusion on Day 1 of each 21-day cycle.
  Other Names: Avastin; RO4876646
  Arms: Cohort A: Atezolizumab+Bevacizumab

SUMMARY:
The purpose of this study is to assess the safety of atezolizumab and bevacizumab, or atezolizumab alone, as first-line treatment in participants with unresectable, locally advanced or metastatic hepatocellular carcinoma (HCC) with Child-pugh B7 or B8 cirrhosis.

DETAILED DESCRIPTION:
This is a Phase II, open-label, multicohort, multicenter study in participants with unresectable, locally advanced, or metastatic HCC who have Child-pugh B7 or B8 liver cirrhosis and have received no prior systemic therapy in this treatment setting. The study is designed to non-comparatively evaluate the safety of atezolizumab plus bevacizumab (Cohort A) or atezolizumab monotherapy (Cohort B) in this population.

ELIGIBILITY:
General Inclusion Criteria:

* Locally advanced or metastatic and/or unresectable HCC with diagnosis confirmed by histology/cytology or clinically by American Association for the Study of Liver Diseases (AASLD) criteria in cirrhotic participants
* Disease that is not amenable to curative surgical and/or locoregional therapies
* No prior systemic treatment (including systemic investigational agents) for locally advanced or metastatic and/or unresectable HCC
* Measurable disease (at least one untreated target lesion) according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 within 7 days prior to initiation of study treatment
* Child-pugh B7 or B8 cirrhosis at screening and within 7 days prior to study treatment
* Adequate hematologic and end-organ function
* Life expectancy of at least 12 weeks
* Female participants of childbearing potential must be willing to avoid pregnancy and egg donation
* Absolute neutrophil count ≥1.0 x 10^9 per liter (/L) (≥1000 per microliter [/μL]) without granulocyte colony-stimulating factor support
* Platelet count ≥ 50 × 109/L (50,000/μL) without transfusion
* Hemoglobin ≥ 80 grams per liter (g/L) (8 grams per deciliter [g/dL]) aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 × upper limit of normal (ULN)
* Serum bilirubin ≤ 3 × ULN
* Creatinine clearance ≥ 50 milliliters per minute (mL/min) (calculated using the Cockcroft-gault formula)
* Serum albumin ≥ 20 g/L (2.0 g/dL) without transfusion in the prior 3 months
* International normalized ratio (INR) ≤2.3

General Exclusion Criteria:

* Pregnancy or breastfeeding
* Prior treatment with cluster of differentiation 137 (CD137) agonists or immune checkpoint blockade therapies
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Treatment with locoregional therapy to liver within 28 days prior to initiation of study treatment, or non-recovery from side effects of any such procedure
* Treatment with systemic immunostimulatory agents
* Treatment with systemic immunosuppressive medication
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment
* Inadequately controlled hypertension
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Participants who have a known concurrent malignancy that is progressing or requires active treatment, who have not completely recovered from treatment, or who have a significant malignancy history that, in the opinion of the investigator, should preclude participation
* Participants on preventative hormonal therapies (i.e., tamoxifen and other hormonal inhibitors) are not excluded
* Known fibrolamellar HCC, sarcomatoid HCC, other rare HCC variant, or mixed cholangiocarcinoma and HCC
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
* Prior allogeneic stem cell or solid organ transplantation
* Actively listed for liver transplantation
* Co-infection with hepatitis B virus (HBV) and hepatitis C virus (HCV)
* Untreated or incompletely treated esophageal and/or gastric varices with bleeding or that are at high risk for bleeding
* A prior bleeding event due to esophageal and/or gastric varices within 6 months prior to initiation of study treatment
* Grade ≥3 hemorrhage or bleeding event within 6 months prior to initiation of study treatment
* Hepatic encephalopathy is allowed if no active symptoms or stable within 3 months of study treatment
* History, planned, or recommended placement of transjugular intrahepatic portosystemic shunt (TIPS) is excluded from Cohort A only. TIPS is acceptable in Cohort B
* Diagnostic paracentesis is allowed. Therapeutic paracentesis: one large volume paracentesis prior to enrollment with diuretic controlled ascites is allowed.
* Participants with ascites controlled on diuretics are allowed
* History of spontaneous bacterial peritonitis within last 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) | Baseline through the end of the study (up to approximately 36 months)
  An AE is any untoward medical occurrence in a participant or clinical study participant temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Severity is determined according to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0) in Cohorts A and B.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (61):
- United States (60):
  - University of Arizona Cancer Center, Tucson, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of Southern California-Keck School of Medicine -1975 Zonal Ave, Los Angeles, California
  - University of Southern California, Newport Beach, California
  - University of California Irvine Medical Center, Orange, California
  - California Liver Research Institute, Pasadena, California
  - University of California Davis Medical Center, Sacramento, California
  - Stanford Health Care, Stanford, California
  - Harbor UCLA Medical Center, Torrance, California
  - Cedars Sinai Comprehensive Transplant Center, West Hollywood, California
  - Rocky Mountain Cancer Centers (Williams) - USOR, Denver, Colorado
  - Hartford Healthcare Cancer Institute at Hartford Hospital, Hartford, Connecticut
  - Washington DC VA Medical Center, Washington D.C., District of Columbia
  - Orlando Health Inc., Orlando, Florida
  - Northwestern University, Chicago, Illinois
  - University of Illinois Health Outpatient Care Center, Chicago, Illinois
  - The Duchossois Center for Advanced Medicine, Chicago, Illinois
  - University of Kentucky - Markey Cancer Center, Lexington, Kentucky
  - LSU Health Baton Rouge, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Veterans Affairs Ann Arbor Healthcare System, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Saint Luke?s Hospital of Kansas City, Kansas City, Missouri
  - MorristownMedicalCenter, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey at University Hospital, Newark, New Jersey
  - Long Island Heart Associates, Mineola, New York
  - R.J. Zuckerberg Cancer Hospital/Northwell Health - BRANY - PPDS, New Hyde Park, New York
  - NYU Langone Medical Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - James J Peters Veterans Administration Medical Center - NAVREF, The Bronx, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Dayton VA Medical Center - NAVREF - PPDS, Dayton, Ohio
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Kaiser Permanente Westside Medical Center, Hillsboro, Oregon
  - OHSU Knight Cancer Institute Hematology Oncology, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Veterans Affairs Pittsburgh Healthcare System - NAVREF - PPDS, Pittsburgh, Pennsylvania
  - The West Clinic (East Campus), Germantown, Tennessee
  - Nashville General Hospital at Meharry, Nashville, Tennessee
  - Liver Institute at Methodist Dallas, Dallas, Texas
  - Moody Outpatient Center ? Parkland Health, Dallas, Texas
  - Texas Oncology (Worth) - USOR, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Oncology - Denison Cancer Center, Denison, Texas
  - Kelsey Research Foundation, Houston, Texas
  - Michael E Debakey VA Medical Center - NAVREF - PPDS, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Intermountain Healthcare, Murray, Utah
  - Intermountain Cancer Center, St. George, Utah
  - Inova Schar Cancer Institute, Falls Church, Virginia
  - Maryview Hospital, Inc., Newport News, Virginia
  - Bon Secours St. Mary's Hospital, Richmond, Virginia
  - VCU Medical Center North Hospital, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
- Pan American Center for Oncology Trials, LLC, Rio Piedras, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing